CLINICAL TRIAL: NCT00697320
Title: Efficacy of NovoSeven® (Activated Recombinant Human Factor VII): Non-interventional Study in Patients With Congenital Haemophilia With Inhibitors, Acquired Haemophilia, Factor FVII Deficiency, and Glanzmann's Thrombasthenia
Brief Title: Observational Study on the Efficacy and Safety of NovoSeven® During "Real-life" Usage in Germany
Acronym: WIRK
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-1921
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Congenital Bleeding Disorder; Congenital FVII Deficiency; Glanzmann's Disease; Acquired Bleeding Disorder; Acquired Haemophilia
MeSH Terms: conditions — Thrombasthenia | interventions — Factor VII; recombinant FVIIa

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — A NON INTERVENTIONAL OBSERVATIONAL STUDY:
  Doses and frequency of injections to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoSeven®; F7; activated recombinant human factor VII

SUMMARY:
This NON INTERVENTIONAL OBSERVATIONAL STUDY is conducted in Europe. The primary aim is to observe the haemostatic efficacy of NovoSeven® treatment during routine practice in German clinics. The observational study observes patients with congenital haemophilia with inhibitors to coagulation factors VIII or IX, acquired haemophilia, congenital FVII deficiency, or Glanzmann's thrombasthenia who have received at least one dose of NovoSeven® for treatment of a bleeding episode or for the prevention of a bleeding when undergoing surgery or an invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from patient or patient's legally acceptable representative in which he agrees that the patient's pseudonymised personal data will be transferred for use in a scientific evaluation and publication

Exclusion Criteria:

* Due to the non-interventional observational character of the study, there are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with congenital haemophilia with inhibitors to coagulation factors VIII or IX, acquired haemophilia, congenital FVII deficiency, or Glanzmann's thrombasthenia who have received at least one dose of NovoSeven®.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of acute bleeding episodes for which haemostasis (defined as stop or significant reduction of bleeding) will be achieved | within 9 hours after initiation of treatment with NovoSeven® or of invasive procedures for which haemostasis will be maintained during the time period of haemostatic coverage with NovoSeven®

SECONDARY OUTCOMES:
Time proportion of acute bleeding treatments resulting in effective pain relief | within 9 hours after initiation of treatment with NovoSeven®
Proportion of patients experiencing one or more re-bleeds | within 24 hours after begin of an acute bleeding episode that was successfully treated with NovoSeven® (stop or significant reduction of bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com